CLINICAL TRIAL: NCT05301426
Title: Differences Between the Effects of the Neural Glide Technique on the Sciatic Nerve and the Passive Stretching Technique in the Short Hamstring Muscles
Brief Title: Neural Glide Technique on the Sciatic Nerve and the Passive Stretching Technique in the Short Hamstring Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Angel Martínez Carrasco, Professor PhD, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FJ-2022-01
Record Dates: First submitted 2022-03-08; First posted 2022-03-29 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Hamstring Muscles; Sciatic Nerve; Flexibility
Keywords: Hamstring muscles; Sciatic nerve; Flexibility

STUDY DESIGN:
Intervention Model Description: Two intervention groups. One control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Masked participants. Masked data analyst.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Passive hamstring stretch. (Experimental): Manual stretching of the hamstring muscles using the technique proposed by Henri Neiger.
  Interventions: Other: Stretching of the hamstring muscles.
- Longitudinal slippage of the sciatic nerve. (Experimental): Neurodynamic technique described by David Butler and Michael Shacklock.
  Interventions: Other: Neural slippage of the sciatic nerve.
- Passive upper limb mobilisations. (Active Comparator): Control group. Passive mobilisation of the upper limbs.
  Interventions: Other: Passive upper limb mobilisations.

INTERVENTIONS:
Other: Stretching of the hamstring muscles. — Passive stretching of the hamstring muscles.
  Arms: Passive hamstring stretch.
Other: Neural slippage of the sciatic nerve. — Neurodynamic technique on the sciatic nerve.
  Arms: Longitudinal slippage of the sciatic nerve.
Other: Passive upper limb mobilisations. — Passive mobilisations performed on the upper limbs used as a placebo.
  Arms: Passive upper limb mobilisations.

SUMMARY:
The project consists of studying the differences between neural gliding techniques of the sciatic nerve and passive stretching of the hamstring muscles in football players.

DETAILED DESCRIPTION:
Study of hamstring shortening in football players through passive muscle stretching and the use of the neurodynamic technique of longitudinal sliding of the sciatic nerve.

ELIGIBILITY:
Inclusion criteria:

* Footballers with shortening of the hamstring musculature.
* Age between 16 and 18 years.
* Subjects who agree to participate in the study.

Exclusion criteria:

* Subjects with significant nerve involvement.
* Subjects with scars or wounds affecting the assessment.
* Subjects with muscle injuries in the lower limb.
* Subjects with herniated discs or chronic acute low back pain.
* Subjects with pain or paresthesia in the lower limbs.

Ages: 16 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Men only.
Enrollment: 50 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Differences between passive stretching of the hamstring muscles and longitudinal sliding of the sciatic nerve. | One month.
  The degree of elasticity of the hamstring musculature will be measured using the Goniometer by placing the hip in 90 degrees flexion and measuring the extension in degrees of the knee.
  A pre-test and post-test measurement will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Martínez Carrasco, PhD, Study Director — Universidad de Murcia
Locations (1):
- Campo de Fútbol de Archena, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No